CLINICAL TRIAL: NCT07060924
Title: Evaluation of Dental Students' Attitudes and Behaviors Toward Intravenous Cannulation: A Comparative Study of Game-Based Learning and Model Arm Practice
Brief Title: Comparison of Game-Based Learning and Model Arm Practice for Teaching Intravenous Cannulation to Dental Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cagil Vural, Associated Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AnkaraU 8/23
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Dental Education and Special Care Dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (GBL Group) (Experimental): Training with 3D Medsim game-based platform for intravenous cannulation before patient application
  Interventions: Behavioral: Game-Based Learning (GBL)
- Arm B (Model Arm Group) (Experimental): Practical training on a circulation model arm for intravenous cannulation before patient application
  Interventions: Behavioral: Model Arm Practice

INTERVENTIONS:
Behavioral: Game-Based Learning (GBL) — Participants in this group received practical training in peripheral intravenous cannulation (PIVC) using a game-based learning (GBL) simulation platform called 3D Medsim. The platform offered a scenario-based training environment that included a structured sequence of pre-test, simulated procedural performance, and post-test. Students were required to perform virtual tasks such as preparing the patient, selecting the correct equipment, identifying the puncture site, and performing cannulation. The simulation provided interactive feedback and scoring. The application was accessible via PC, tablet, or smartphone, allowing students to practice flexibly. Training was conducted under the supervision of an anesthesiologist.
  Arms: Arm A (GBL Group)
Behavioral: Model Arm Practice — Participants in this group practiced PIVC using a high-fidelity model arm simulator designed to replicate human anatomy and venous access. The training model included artificial veins (basilic, cephalic, median cubital, and metacarpal) with realistic skin layers and a circulation system that mimicked blood flow. Students practiced cannulation techniques including vein localization, needle insertion, and catheter placement. The hands-on training provided tactile and visual feedback, and all procedures were supervised by an anesthesiologist. This method aimed to develop psychomotor skills and confidence through realistic simulation.
  Arms: Arm B (Model Arm Group)

SUMMARY:
This randomized controlled study aimed to compare the effectiveness of game-based learning (GBL) and model arm practice in teaching peripheral intravenous cannulation (PIVC) skills to final-year dental students. Sixty participants were randomly assigned to two groups. The impact of each method was assessed in terms of procedural success, anxiety levels (STAI), self-confidence (VAS), and student satisfaction.

DETAILED DESCRIPTION:
Peripheral intravenous cannulation (PIVC) is a complex procedure now integrated into the Turkish National Dental Curriculum (DUÇEP). This study compared the effectiveness of GBL using the 3D Medsim platform and model arm practice in training students on PIVC. Participants were final-year dental students with no prior PIVC experience. Pre- and post-intervention evaluations included procedural success (simulation or model), anxiety (STAI), self-confidence (VAS), and satisfaction (Likert scale). Clinical success was also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Final-year dental students at Ankara University
* No prior experience with PIVC
* Volunteered and provided informed consent

Exclusion Criteria:

* Any prior practical experience in intravenous cannulation
* Refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Procedural Success Rate in Clinical Application | Within 1 week after training
  The rate of successful intravenous cannulation performed by students on real patients under supervision. Success was defined as a successful puncture and catheter placement on the first or second attempt. Assessed by an anesthesiologist during clinical practice.
Change in Self-Confidence Level (VAS Score) | From pre-training to post-clinical application (within 2 weeks)
  Students marked their perceived self-confidence regarding PIVC on a 10-cm visual analog scale (0 = no confidence, 10 = full confidence). Measurements were taken both after training and after clinical application.

SECONDARY OUTCOMES:
Change in State Anxiety Level (State-Trait Anxiety Inventory - State Scale) | Baseline (pre-training), immediately after training, and immediately after clinical application (all within 2 weeks)
  Anxiety was measured using the State-Trait Anxiety Inventory - State Scale (STAI-S), a validated 20-item questionnaire assessing situational anxiety. Each item is rated on a 4-point Likert scale, yielding total scores ranging from 20 to 80, where higher scores indicate higher levels of anxiety (i.e., a worse psychological outcome).
Satisfaction with Training Method (Likert Questionnaire) | Immediately after training
  A 5-item satisfaction questionnaire evaluated participants' perceptions of the training method's usefulness, content diversity, presentation, motivation, and compatibility with learning style. Each item was scored on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Dentistry, Ankara, Turkey (Türkiye)